CLINICAL TRIAL: NCT05408299
Title: Comparative Study of Patterns of Immune Response to COVID 19 Vaccination Between Immunocompetent and Immunocompromised Subjects
Brief Title: Comparative Study of Patterns of Immune Response to COVID 19 Vaccination
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Research Centre, Egypt (Other)
Collaborators: The holding company for biological products and vaccines (VACSERA) (Unknown); Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Mohamed Aly Abd El Salam Mokhles, Professor of Gastroenterology and Hepatology, National Research Centre, Egypt
Other Study IDs: 03/22-0001
Record Dates: First submitted 2022-06-05; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Immune Response to Covid 19 Vaccination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immunocompetent: 100 healthy persons not suffering of any systemic diseases or malignancy of whatever nature.
  Interventions: Biological: Covid vaccines (Moderna - Pfizer- Astra Zeneca- Johnson and Johnson - Sinopahrm)
- Immunocompromised: 100 B thalassemia splenectomised patients.
  Interventions: Biological: Covid vaccines (Moderna - Pfizer- Astra Zeneca- Johnson and Johnson - Sinopahrm)

INTERVENTIONS:
Biological: Covid vaccines (Moderna - Pfizer- Astra Zeneca- Johnson and Johnson - Sinopahrm) — Vaccination

SUMMARY:
An effective vaccine stands as the most effective way for controlling the COVID 19 pandemic , yet, immunogenic vaccine efficacy needs to be extensively studied . T cell responses against the structural proteins have been found to be the most immunogenic in peripheral blood mononuclear cells of convalescent SARS-CoV1 patients which needs to be tested in SARS -COV2 vaccine efficacy studies alongside with the sustainability of humoral and cellular immune responses . Clinically , immunocompromised patients face drastic outcome of infections , which led the Advisory Committee on Immunization Practices (ACIP) - USA -and the Joint Committee on Vaccination and Immunisation (JCVI) -UK- recommend COVID-19 vaccination of immunocompromised , the WHO Strategic Advisory Group of Experts on Immunization (SAGE), recommended that the three vaccines(Pfizer ,Moderna and Astra Zeneca) can be used for individuals with high-risk comorbidities . Nevertheless, there is an unmet research need concerning the immune response towards COVID 19 vaccination in this population .

Based on the previous work of our team in designing B and T cell epitopes distributed over the S protein , we will study the immune response in the available vaccines in Egypt.

DETAILED DESCRIPTION:
This proposed project is a joint collaboration between the National Research Center(NRC) , Hematology treatment unit of the holding company for biological products and vaccines (VACSERA) and Theodor Bilharz research institute . After a 1 month period of preparation , enrollment will start at month 2 (M2) over a 2 months enrollment window, where persons from 18-70 years old , of both sexes , having their first vaccination dose no more than 3 weeks of any of the available vaccines in Egypt will be enrolled into the project after signing an informed consent . Healthy persons not suffering from any systemic diseases will be enrolled from Theodor Bilharz vaccination center , and the Medical Researches Center of Excellence ( MRCE) at the NRC from the NRC vaccinated staff , while splenectomised B thalassemia patients will be enrolled from the hematology treatment unit at VACSERA . First visit will be performed 3 weeks post the first vaccination dose , while the second visit will be performed 3 weeks post the second vaccination dose , and the third visit will be performed 3 months post the second vaccination dose where ( 5 ) ml of blood will be withdrawn at each visit for the determination of the primary immune response at the first 2 visits and the sustainability of the immune response at the third visit . Enrolled persons will be instructed to contact the project logistics administrator upon experiencing any suspicious symptom of COVID 19 infection ( Fever- loss of taste and/or smell - myalgia - malaise - headache - diarrhea ) who will arrange for an additional visit where a PCR test for COVID 19 will be performed for the determination of breakthrough infections , and if positive this will be considered a primary end point and an additional ( 5) ml of blood will be withdrawn for testing for the immune status .

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes.
2. 3 weeks post scheduled first vaccination dose
3. Healthy group not suffering from any systemic diseases.
4. B thalassemia major splenectomized group
5. Signing an informed consent .

Exclusion Criteria:

1- Malignancy of whatever nature. 2- Systemic diseases apart from B thalassemia for the B thalassemia group. 3- Previous infection with COVID 19 . 4- Refusal to sign the informed consent .

-

Ages: 15 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study will comprise 200 subjects divided into 2 groups; Group 1 : 100 healthy subjects not suffering of systemic diseases vaccinated at any of the MOH vaccination centers. Group 2: 100 B thalssemia splenectomised patients representing an immunocompromised cohort.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-20 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Studying the immune response to COVID -19 vaccination | Month 3-Month 9 of the study
  Detection of total induced IgG binding antibodies
. Comparing immune response to COVID 19 vaccination between healthy and immunocompromised groups | Month 3 - Month 9 of the study

SECONDARY OUTCOMES:
. Determination of the most immunogenic parts of COVID 19 vaccine | Month 3-Month 9 of the study
  Detecting the most immunogenic epitopes located within the spike protein of the vaccines through ELispot assay

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Mokhles, Professor, Principal Investigator — National Research Center .
Locations (1):
- National Research Center, Cairo, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through published scientific papers that come out of the study , in addition to conferences presentations.
Supporting Information: Study Protocol, SAP
Time Frame: AT month 12 of the study